CLINICAL TRIAL: NCT01939964
Title: A Double-Blind, Randomized, Placebo-controlled Study to Compare the Efficacy and Safety of Rena ™ Activation Mist on Facial Skin Wrinkles.
Brief Title: Study to Determine Effectiveness of Activation Mist on Facial Skin Wrinkles
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: California Allergy and Asthma Medical Group, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0012
Record Dates: First submitted 2013-09-07; First posted 2013-09-11 (Estimated); Last update posted 2013-09-11 (Estimated); Status verified 2013-09

CONDITIONS: Skin Wrinkles on Face and Neck Areas
Keywords: Wrinkles; Activation Mist

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Activation Mist (Active Comparator): Liquid mist preparation to be sprayed topically on wrinkle areas
  Interventions: Other: Activation Mist
- Placebo (Placebo Comparator): sugar pill
  Interventions: Other: Activation Mist

INTERVENTIONS:
Other: Activation Mist — Activation Mist topical spray
  Other Names: AM

SUMMARY:
To determine the effect of Activation Mist (AM) on skin wrinkles and appearance.

DETAILED DESCRIPTION:
This study aims to study the effects of Activation Mist ( AM) on skin wrinkles. It contains a proprietary blend of minerals and nutritional supplements which is patented as "Liquidized Infrared Negative Ion Activation Energy". Active ingredients include sodium bicarbonate, potassium bicarbonate, sodium carbonate, strontium carbonate, gold nanoparticles, calcium, germanium, selenium , zinc, sugar and water. When applied to the skin , it has been shown to reduce the appearance of wrinkles by stimulation of skin fibroblasts to produce new collagen while removing aging dermis cells, facilitate the production of fibrillin proteins and protect the skin from ultraviolet rays.

ELIGIBILITY:
Inclusion Criteria:

1.Male and female subjects aged 30 to 80 years of age with significant facial wrinkles as assessed by the study physician.

Exclusion Criteria:

1. Women who are pregnant or lactating.
2. Subjects with skin conditions that are deemed by the investigator to interfere with the results of this study , including but not limited to: uncontrolled acne, rosacea, atopic dermatitis.
3. Subjects with clinically significant cardiovascular, neurological, renal, endocrine or hematological abnormalities uncontrolled on current therapy.
4. Subjects with history of skin malignancy
5. Subjects with signs of recent sunburn
6. Use of any of the following medications, within 1 week specified of visit 1

   1. Systemic steroids
   2. Topical steroids used on the face
   3. Topical facial preparations including but not limited to: salicylic acid and other acne products, tacrolimus, pimecrolimus.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-11; Primary Completion 2014-06 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Silicone skin replica analysis | before and after 8 weeks of treatment
  Silflo ™ vinyl silicone ( Cuderm Corp.) is applied to the skin areas to be studied and replicas obtained after letting it stand for 3- 5 minutes. The replica technique takes a negative copy of the skin surface which is analyzed by optical profilometry. Optical profilometry ( BioNet Inc.) uses light intensity to assess skin wrinkle texture by objective parameters ( e.g. spacing, breadth, shadows, num wrinkles) This will be performed before and after 8 weeks of treatment.

SECONDARY OUTCOMES:
Wrinkle Score | every week for 8 weeks
  A blinded evaluation will assess wrinkle appearance and grade on a scale of 0 to 5
Photographic evaluation | weekly for 8 weeks
  A blinded evaluator will assess photographs of wrinkles and evaluate presence or absence of improvement

CONTACTS AND LOCATIONS:
Locations (1):
- California Allergy and Asthma Medical Group, Los Angeles, California, United States

REFERENCES:
- See also: Research site website — http://www.calallergy.com